CLINICAL TRIAL: NCT00473941
Title: Expressive Writing and Adjustment to Colorectal Cancer
Brief Title: Life After Cancer: Behavioral Treatment Study to Improve Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R21CA107428-01A2 (NIH)
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Writing in a journal 15 minutes a day
  Interventions: Behavioral: Expressive writing
- 2 (Placebo Comparator): Control Writing in a journal 15 minutes a day
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Expressive writing — Behavioral intervention using writing about cancer to improve quality of life outcomes

SUMMARY:
The purpose of the study is to find new ways to improve the quality of life of people who have been treated for colon or rectal cancer.

DETAILED DESCRIPTION:
Individuals who take part in the study can expect:

Two Interviews:

* To be interviewed by our research staff over the phone. The interviews will include questions about your current quality of life and health.

Brief Writing in a Journal:

* To write for 15 minutes twice a week for two weeks about aspects of your life.

ELIGIBILITY:
Inclusion Criteria:

* Treated for stage I, II or III colon or rectal cancer in the past 5 years
* Completed surgical treatment
* Must be able to read and write in English

Exclusion Criteria:

* History of other cancers, with the exception of non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 2-Weeks
  self-report depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lepore, Ph.D., Principal Investigator — Temple University; Tracey A Revenson, Ph.D, Principal Investigator — Graduate College, City University of New York
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Colon Cancer Alliance — http://www.ccalliance.org/
- See also: Cancer Information Network — http://www.cancerlinksusa.com/colorectal/index.asp